CLINICAL TRIAL: NCT06091397
Title: Validation of the Italian Version of the Forgotten Joint Score (FJS-12) as a Patient-reported Outcome Measure in Total Ankle Replacement: a Study on an Italian Population
Brief Title: Validation of the Italian Version of the Forgotten Joint Score (FJS-12) in Total Ankle Replacement
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Antonio Mazzotti, Principal Investigator, Istituto Ortopedico Rizzoli
Other Study IDs: FORG-Score
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: PROMs; Total Ankle Replacement; Italian Forgotten Joint Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The arthritic pathology of the tibio-tarsal joint has a prevalence of approximately 1% in the general population, and its incidence has been increasing over the years. Advanced-stage arthritis causes pain, impairs mobility, and has an extremely negative impact on patients' quality of life, resulting in significant social and economic costs. Unlike hip and knee arthritis, ankle arthritis is often secondary to traumatic events, affecting younger patients. An emerging treatment for severe ankle arthritis is ankle prosthetic replacement, and patient-reported outcome measures (PROMs) are increasingly used to assess patient outcomes. The study focuses on the validity and reproducibility of the Italian versione of the Forgotten Joint Score (FJS) in ankle prostheses, obtained through the translation-back-translation method, with a sample size of 120 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either gender, aged between 25 and 80 years;
* Patients who have undergone total ankle replacement surgery for tibio-tarsal joint pathology starting from 2018, as well as new patients on the waiting list.
* Signed informed consent for participation in the study;
* Patients who are prepared and motivated to attend the scheduled follow-up visits and complete the study questionnaires.

Exclusion Criteria:

* Patients unable to understand or consent;
* BMI > 40.
* Refusal to complete the study consent form.
* Substance abuse or psychological disorders that could interfere with the ability to comply with rehabilitation programs and postoperative assessments.
* Known sensitivity to device materials.
* Presence of an active or suspected latent infection in or around the affected ankle joint.

Ages: 25 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients aged between 25 and 80 years, suffering from degenerative pathology of the tibio-tarsal joint, who have undergone surgical total ankle prosthetic replacement.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
IFJS - Italian Forgotten Join Score | At baseline (day 0)
  The Italian Forgotten Joint Score (FJS) is the italian versione of the Forgotten Joint score that is a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. 0 worst possible score, 100 best possible score
IFJS - Italian Forgotten Join Score | After 3 months
  The Italian Forgotten Joint Score (FJS) is the italian versione of the Forgotten Joint score that is a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. 0 worst possible score, 100 best possible score
IFJS - Italian Forgotten Join Score | After 6 months
  The Italian Forgotten Joint Score (FJS) is the italian versione of the Forgotten Joint score that is a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. 0 worst possible score, 100 best possible score
IFJS - Italian Forgotten Join Score | After 12 months
  The Italian Forgotten Joint Score (FJS) is the italian versione of the Forgotten Joint score that is a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. 0 worst possible score, 100 best possible score
IFJS - Italian Forgotten Join Score | After 24 months
  The Italian Forgotten Joint Score (FJS) is the italian versione of the Forgotten Joint score that is a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. 0 worst possible score, 100 best possible score
IFJS - Italian Forgotten Join Score | After 36 months
  The Italian Forgotten Joint Score (FJS) is the italian versione of the Forgotten Joint score that is a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. 0 worst possible score, 100 best possible score
IFJS - Italian Forgotten Join Score | After 48 months
  The Italian Forgotten Joint Score (FJS) is the italian versione of the Forgotten Joint score that is a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. 0 worst possible score, 100 best possible score
IFJS - Italian Forgotten Join Score | After 60 months
  The Italian Forgotten Joint Score (FJS) is the italian versione of the Forgotten Joint score that is a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint. Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score. 0 worst possible score, 100 best possible score

SECONDARY OUTCOMES:
American Orthopedic Foot and Ankle Society (AOFAS score) | At baseline (day 0)
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
American Orthopedic Foot and Ankle Society (AOFAS score) | After 3 months
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
American Orthopedic Foot and Ankle Society (AOFAS score) | After 6 months
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
American Orthopedic Foot and Ankle Society (AOFAS score) | After 12 months
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
American Orthopedic Foot and Ankle Society (AOFAS score) | After 24 months
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
American Orthopedic Foot and Ankle Society (AOFAS score) | After 36 months
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
American Orthopedic Foot and Ankle Society (AOFAS score) | After 48 months
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
American Orthopedic Foot and Ankle Society (AOFAS score) | After 60 months
  The American Orthopedic Foot and Ankle Society Score is a semi-objective rating scale that evaluates ankle pain, motion and alignment and ranges from 0 to 100 points. 0 worst possible score, 100 best possible score
MOXFQ (Manchester-Oxford Foot Questionnaire) | At baseline (day 0)
  The MOXFQ is a 16-item instrument answered on a five-point Likert scale (each item is scored from 0 to 4, with 4 denoting 'most severe'). Scores for each item are summed to form three separate subscales representing underlying domains: walking/standing problems (seven items), foot pain (five items), and issues related to social interaction (four items). Raw scale scores are then each converted to a metric from 0 to 100, where 100 denotes the most severe.
MOXFQ (Manchester-Oxford Foot Questionnaire) | After 3 months
  The MOXFQ is a 16-item instrument answered on a five-point Likert scale (each item is scored from 0 to 4, with 4 denoting 'most severe'). Scores for each item are summed to form three separate subscales representing underlying domains: walking/standing problems (seven items), foot pain (five items), and issues related to social interaction (four items). Raw scale scores are then each converted to a metric from 0 to 100, where 100 denotes the most severe.
MOXFQ (Manchester-Oxford Foot Questionnaire) | After 6 months
  The MOXFQ is a 16-item instrument answered on a five-point Likert scale (each item is scored from 0 to 4, with 4 denoting 'most severe'). Scores for each item are summed to form three separate subscales representing underlying domains: walking/standing problems (seven items), foot pain (five items), and issues related to social interaction (four items). Raw scale scores are then each converted to a metric from 0 to 100, where 100 denotes the most severe.
MOXFQ (Manchester-Oxford Foot Questionnaire) | After 12 months
  The MOXFQ is a 16-item instrument answered on a five-point Likert scale (each item is scored from 0 to 4, with 4 denoting 'most severe'). Scores for each item are summed to form three separate subscales representing underlying domains: walking/standing problems (seven items), foot pain (five items), and issues related to social interaction (four items). Raw scale scores are then each converted to a metric from 0 to 100, where 100 denotes the most severe.
MOXFQ (Manchester-Oxford Foot Questionnaire) | After 24 months
  The MOXFQ is a 16-item instrument answered on a five-point Likert scale (each item is scored from 0 to 4, with 4 denoting 'most severe'). Scores for each item are summed to form three separate subscales representing underlying domains: walking/standing problems (seven items), foot pain (five items), and issues related to social interaction (four items). Raw scale scores are then each converted to a metric from 0 to 100, where 100 denotes the most severe.
MOXFQ (Manchester-Oxford Foot Questionnaire) | After 36 months
  The MOXFQ is a 16-item instrument answered on a five-point Likert scale (each item is scored from 0 to 4, with 4 denoting 'most severe'). Scores for each item are summed to form three separate subscales representing underlying domains: walking/standing problems (seven items), foot pain (five items), and issues related to social interaction (four items). Raw scale scores are then each converted to a metric from 0 to 100, where 100 denotes the most severe.
MOXFQ (Manchester-Oxford Foot Questionnaire) | After 48 months
  The MOXFQ is a 16-item instrument answered on a five-point Likert scale (each item is scored from 0 to 4, with 4 denoting 'most severe'). Scores for each item are summed to form three separate subscales representing underlying domains: walking/standing problems (seven items), foot pain (five items), and issues related to social interaction (four items). Raw scale scores are then each converted to a metric from 0 to 100, where 100 denotes the most severe.
MOXFQ (Manchester-Oxford Foot Questionnaire) | After 60 months
  The MOXFQ is a 16-item instrument answered on a five-point Likert scale (each item is scored from 0 to 4, with 4 denoting 'most severe'). Scores for each item are summed to form three separate subscales representing underlying domains: walking/standing problems (seven items), foot pain (five items), and issues related to social interaction (four items). Raw scale scores are then each converted to a metric from 0 to 100, where 100 denotes the most severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Matsumoto M, Baba T, Homma Y, Kobayashi H, Ochi H, Yuasa T, Behrend H, Kaneko K. Validation study of the Forgotten Joint Score-12 as a universal patient-reported outcome measure. Eur J Orthop Surg Traumatol. 2015 Oct;25(7):1141-5. doi: 10.1007/s00590-015-1660-z. Epub 2015 Jul 7. PMID 26148699